CLINICAL TRIAL: NCT06045780
Title: Study on the Mechanism of Endotoxic Acute Lung Injury-induced Golgi Stress Based on Regulating HO-1/CREB3
Brief Title: HO-1/CREB3 Modulates Golgi Stress in Patients With Sepsis
Status: Recruiting | Type: Observational
Sponsor: Tianjin Nankai Hospital (Other)
Responsible Party: Principal Investigator, Jianbo Yu, Prof., Tianjin Nankai Hospital
Other Study IDs: NKYY_YXKT_IRB_2023_049_01
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The peripheral blood mononuclear cells (PBMCs) were acquired from blood by a density gradient centrifugation method (Ficoll Histopaque); peripheral blood of normal subjects and septic cases.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis: disease
  Interventions: Other: nothing
- Healthy controls: healthy
  Interventions: Other: nothing

INTERVENTIONS:
Other: nothing — disease

SUMMARY:
This study was an ambispective observational cohort study that included sepsis patients hospitalized in the Intensive care unit (ICU) of the Nankai Hospital. All patients met the consensus criteria of sepsis-3. The purpose of this study is to investigate the valuable biomarkers for the severity of sepsis and predictors of 30-day mortality for patients with sepsis.

DETAILED DESCRIPTION:
All patients met the consensus criteria of sepsis-3. The purpose of this study is to investigate the valuable biomarkers for the severity of sepsis and predictors of 30-day mortality for patients with sepsis.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females over the age of 18;
2. Sepsis was diagnosed within 48h which meets SPESIS 3 criteria;
3. Capable of understanding the purpose and risk of the study;
4. Patients or proxy must give written informed consent before any assessment is performed.

Exclusion Criteria:

1. Pregnancy, lactation or perinatal period;
2. Breast carcinoma;
3. HIV seropositive or Syphilis seropositive;
4. Any clinical-relevant condition that might affect study participation and/or study results;
5. Participation in any other intervention trial;
6. Unwillingness or inability to following the study protocol in the investigators opinion.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Septic patients and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
cAMP-response element binding protein 3, CREB3 | Up to Day 28
  CREB3 levels were measured in the PBMCs of sepsis patients and healthy controls
ADP-ribosylation factor 4, ARF4 | Up to Day 28
  ARF4 levels were measured in the PBMCs of sepsis patients and healthy controls

SECONDARY OUTCOMES:
Heme oxygnase-1, HO-1 | Up to Day 28
  HO-1 levels were measured in the PBMCs of sepsis patients and healthy controls
ARF family | Up to Day 28
  ARF1, ARF3, ARF5, ARF6 levels were measured in the PBMCs of sepsis patients and healthy controls
Oxygenation index | Up to Day 28
  The ratio of arterial oxygen partial pressure (PaO2 in mmHg) to fractional inspired oxygen (FiO2 expressed as a fraction, not a percentage).
Mechanical ventilation days | Up to Day 28
  The number of days the patient was alive and mechanical ventilating
Inflammation biomarkers Inflammation levels | Up to Day 28
  Procalcitonin (PCT), C-reactive protein (CRP), tumor necrosis factor-alpha (TNF-alpha), interleukin-1 beta (IL-1β), and interleukin-6 (IL-6)
ICU stay length | Up to Day 90
  The number of days the patient was alive and ICU stay
28 days survive | Up to Day 28
  All Cause Mortality to Day 28
Sequential Organ-Failure Assessment (SOFA) score | Up to Day 28
  The SOFA score is used to assess the severity and prognosis of sepsis. SOFA was based on six different scores, one for each of the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems each scored from 0 to 4 with an increasing score reflecting worsening organ dysfunction.
Acute Physiology and Chronic Health Evaluation II (APACHE II) score | Up to Day 28
  The APACHE II score consists of three parts: acute physiological score, age score, and chronic health score. APACHE II uses a point score (range 0 to 71) based upon initial values of 12 routine physiologic measurements, age, and previous health status to provide a general measure of severity of disease, with an increasing score reflecting worsening organ dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Jianbo Yu, MD, Study Director — Tianjin Nankai Hospital
Locations (1):
- Tianjin Nankai Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fowler AA 3rd, Truwit JD, Hite RD, Morris PE, DeWilde C, Priday A, Fisher B, Thacker LR 2nd, Natarajan R, Brophy DF, Sculthorpe R, Nanchal R, Syed A, Sturgill J, Martin GS, Sevransky J, Kashiouris M, Hamman S, Egan KF, Hastings A, Spencer W, Tench S, Mehkri O, Bindas J, Duggal A, Graf J, Zellner S, Yanny L, McPolin C, Hollrith T, Kramer D, Ojielo C, Damm T, Cassity E, Wieliczko A, Halquist M. Effect of Vitamin C Infusion on Organ Failure and Biomarkers of Inflammation and Vascular Injury in Patients With Sepsis and Severe Acute Respiratory Failure: The CITRIS-ALI Randomized Clinical Trial. JAMA. 2019 Oct 1;322(13):1261-1270. doi: 10.1001/jama.2019.11825. PMID 31573637